CLINICAL TRIAL: NCT04460092
Title: The Effect of Using 32 - Gauge Needles With Lengths of 5 mm and 8 mm on Pain Post-injection, Leak and Blood Glucose Control in Type - II Diabetic Patients in Baqiyatollah Hospital and Clinic, Tehran, 2019 -2020
Brief Title: Using 32 - Gauge Needles With Lengths of 5 mm and 8 mm on Pain Post-injection, Leak and Blood Glucose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IR.BMSU.BAQ.REC.1398.059
Record Dates: First submitted 2020-05-10; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Blood Glucose; Pain; leakage; insulin injections
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pain | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "A" (Experimental): In the first three days, participants in group "A" will inject 90-degree insulin injections using 5-mm 32-gauge needles. Then, with an interval of one day, in the second three days, they will use 32-gauge needles with a length of 8 mm to inject insulin.
  Interventions: Device: 5-mm 32-gauge Insulin needles in the first three days of Intervention; Device: 8-mm 32-gauge Insulin needles in the last three days of Intervention
- Group"B" (Experimental): In the first three days, participants in group "B" will inject 90-degree insulin injections using 8-mm 32-gauge needles. Then, with an interval of one day, in the second three days, they will use 32-gauge needles with a length of 5mm to inject insulin.
  Interventions: Device: 8-mm 32-gauge Insulin needles in the first three days of Intervention; Device: 5-mm 32-gauge Insulin needles in the last three days of Intervention

INTERVENTIONS:
Device: 5-mm 32-gauge Insulin needles in the first three days of Intervention — 32-gauge needles with a length of 5mm to inject insulin in first three days
  Arms: Group "A"
Device: 8-mm 32-gauge Insulin needles in the first three days of Intervention — 32-gauge needles with a length of 8mm to inject insulin in first three days
  Arms: Group"B"
Device: 5-mm 32-gauge Insulin needles in the last three days of Intervention — 32-gauge needles with a length of 5mm to inject insulin in second three days
  Arms: Group"B"
Device: 8-mm 32-gauge Insulin needles in the last three days of Intervention — 32-gauge needles with a length of 8mm to inject insulin in second three days
  Arms: Group "A"

SUMMARY:
This is a Clinical crossover trial study. In this study, 100 patients with type II diabetes will be selected based on entry and exit criteria, then randomly divided into two equal groups (group "A" and group "B").In the first three days of the first week of hospitalization, in group "A" insulin injection with a 90-degree angle and using Nidel 32-Gauge with a length of 5 mm, and in the other group insulin injection with a 90-degree angle and using Nidel 32-Gauge with a length of 8 mm will be done. After a one-day break, in another three days, the types of needles used in the two groups are moved together. After a one-day break, in another three days, the types of needles used in the two groups are replaced together. Then the VAS scale will be used to assess post-injection pain; the amount of leakage after the injection will be measured in two ways Yes/No, according to the researcher's observation. And to check the effect of Needles on controlling patients' blood sugar, their blood sugar levels will be measured based on the routine of hospital units.

DETAILED DESCRIPTION:
This is a Clinical crossover trial study. In this study, 100 patients with type II diabetes will be selected based on entry and exit criteria, then randomly divided into two equal groups (group "A" and group "B").In the first three days of the first week of hospitalization, in group "A" insulin injection with a 90-degree angle and using Nidel 32-Gauge with a length of 5 mm, and in the other group insulin injection with a 90-degree angle and using Nidel 32-Gauge with a length of 8 mm will be done. After a one-day break, in another three days, the types of needles used in the two groups are moved together. After a one-day break, in another three days, the types of needles used in the two groups are replaced together. Then the VAS scale will be used to assess post-injection pain; the amount of leakage after the injection will be measured in two ways Yes/No, according to the researcher's observation. And to check the effect of Needles on controlling patients' blood sugar, their blood sugar levels will be measured based on the routine of hospital units.

After entering the data in SPSS20 software, the collected data will be analyzed using descriptive statistics (frequency, percentage, mean, standard deviation) and statistical tests (t-test, chi-square).

ELIGIBILITY:
Inclusion Criteria:

* Having type II diabetes
* Use injectable insulin for at least two years
* BMI >18
* Lack of mental illness and mental retardation
* Use insulin pen

Exclusion Criteria:

* Lack of desire to participate in the study
* Having a skin problem in the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-29 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | Up to 7 days
  Laboratory check the Plasma glucose according to the routine of the hospital units
Insulin leakage | Up to 7 days
  The rate of insulin leakage after injection is observational
Pain when insulin injection | Up to 7 days
  Survey severity pain when insulin injection by Visual Analogue Scale (VAS). This is a numerical scale that tells the patient the severity of their pain from one to ten. The larger the number, the more pain there is.

CONTACTS AND LOCATIONS:
Overall Officials: Esmail Heidaranlu, Study Chair — Baqiyatallah Medical Sciences University
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran